CLINICAL TRIAL: NCT04956822
Title: Application of Motor Unit Estimation Index in Amyotrophic Lateral Sclerosis and Related Diseases
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: M2018223
Record Dates: First submitted 2021-06-27; First posted 2021-07-09 (Actual); Last update posted 2021-07-09 (Actual); Status verified 2021-06

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- ALS: Amyotrophic lateral sclerosis group
  Interventions: Other: Basic information; Other: Functional scores; Device: MINUX
- CMT: peroneal muscular dystrophy group
  Interventions: Other: Basic information; Other: Functional scores; Device: MINUX
- KD: Kennedy's disease group
  Interventions: Other: Basic information; Other: Functional scores; Device: MINUX
- Control: Healthy control group
  Interventions: Other: Basic information; Other: Functional scores; Device: MINUX

INTERVENTIONS:
Other: Basic information — Demographic data registration, medical history taking, physical examination. Electrocardiogram. Pulmonary function tests.
Other: Functional scores — depending on the diseases enrolled, ALS and KD chose ALS-FRS functional scores and CMT chose CMTNS2 functional scores
Device: MINUX — MUNIX examination was performed on all subjects. A total of eight bilaterally symmetrical muscles were selected, bilateral abductor little finger or abductor pollicis brevis, bilateral biceps or deltoid muscles, bilateral tibialis anterior muscles, and bilateral femurs. For quadriceps, choose a muscle with less muscle atrophy.

SUMMARY:
This was a cross-sectional study in which patients were divided into 20 patients with amyotrophic lateral sclerosis, 20 patients with peroneal muscular dystrophy, 20 patients with Kennedy's disease and 30 healthy controls, in which patients with amyotrophic lateral sclerosis continued to be followed up for 1 year and the results of 4 cross-sectional examinations were taken.

DETAILED DESCRIPTION:
Background Amyotrophic lateral sclerosis (ALS) is a neurodegenerative disease that usually starts in middle age and manifests mainly as progressive atrophy and weakness of skeletal muscles throughout the body, with death from respiratory muscle involvement after 3 to 5 years. There are no biomarkers for early diagnosis and no effective treatments. Because of the rapid progression of amyotrophic lateral sclerosis, it is important to find indicators that can objectively reflect early changes in the disease. The motor unit number index (MUNIX) is a non-invasive, rapid and objective method to assess the number of motor units, which reflects the loss of motor neurons and has its theoretical basis in monitoring early disease progression.

Objective To explore the diagnostic value of MUNIX in motor neuron disease and other related disorders.

To investigate the role of the 1-year rate of change of MUNIX in monitoring the disease progression in patients with amyotrophic lateral sclerosis.

To investigate the role of MUNIX in predicting survival analysis of ALS patients

[Design] This was a cross-sectional study in which patients were divided into 20 patients with amyotrophic lateral sclerosis, 20 patients with peroneal muscular dystrophy, 20 patients with Kennedy's disease and 30 healthy controls, in which patients with amyotrophic lateral sclerosis continued to be followed up for 1 year and the results of 4 cross-sectional examinations were taken.

ELIGIBILITY:
Inclusion Criteria:

* ALS patient group: 20 patients with confirmed or proposed ALS meeting the 1998 revised El Escorial diagnostic criteria for limb onset ALS.
* CMT group: 20 patients with peroneal muscular dystrophy meeting the genetically confirmed diagnosis, who signed an informed consent form.
* KD group: 20 patients with genetically confirmed Kennedy's disease consistent with genetic diagnosis, signed informed consent.
* healthy controls:

  1. age-matched healthy adults who volunteered to participate;
  2. definite exclusion of tremor, tonicity, and prior brain disease;
  3. exclusion of common disorders affecting peripheral nerves such as entrapment peripheral neuropathy, diabetic peripheral neuropathy, and alcoholic peripheral neuropathy;
  4. signed informed consent.

Exclusion Criteria:

1. signs of sensory impairment;
2. significant sphincter dysfunction;
3. visual and oculomotor impairment;
4. autonomic dysfunction;
5. signs of extravertebral symptoms;
6. severe cortical dysfunction;
7. ALS-like syndrome.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: ALS is a degenerative disease of the nervous system, with an incidence of 2-3 in 100,000. It usually begins in middle age and mainly presents with progressive atrophy and weakness of skeletal muscles throughout the body. After 3 to 5 years, it dies of respiratory muscle involvement. At present, there are no biomarkers for early diagnosis and no effective treatment.
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
The number of motor unit | 1 year
  Motor unit estimation index (MUNIX) is a non-invasive electrophysiological technique that uses compound muscle action potential (CMAP) and surface electromyographic interference pattern (SIP) methods to evaluate the number of motor units (Mus) (motor unit number size, MUSIX).
The size of motor unit | 1 year
  Motor unit estimation index (MUNIX) is a non-invasive electrophysiological technique that uses compound muscle action potential (CMAP) and surface electromyographic interference pattern (SIP) methods to evaluate the number and size of motor units (Mus) (motor unit number size, MUSIX).

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoxuan Liu, Principal Investigator — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No